CLINICAL TRIAL: NCT03102086
Title: The Association Between Nephrolithiasis and Periodontal Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, machtei, Prof, Rambam Health Care Campus
Other Study IDs: 0097-16-RMB
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-03

CONDITIONS: Periodontal Diseases; Nephrolithiasis
MeSH Terms: conditions — Periodontal Diseases; Nephrolithiasis | interventions — Tooth Exfoliation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — kidney stones and dental calculus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Scaling — Scaling of dental calculus

SUMMARY:
Dental calculus is a calcified deposits firmly attached to teeth and implants surfaces. Dental calculus is strongly associated with periodontitis and considered to have indirect role in the pathogenesis of periodontal diseases. Dental calculus composed primarily of calcium phosphate mineral salts originated in the saliva covered by unmineralized bacterial layer. Composition of calculus varies from person to person and influenced by numerous variables such as: age, gender systemic disease and ethnic background.

Nephrolithiasis (kidney stones) are composed of insoluble salts of constituents of the forming urine. The most two frequent stone types are: Calcium oxalate (with a frequency of 15% -35%) and Calcium phosphate (5% -20%). The prevalence of kidney stones varies with race, sex, and geographic location. In the United States for men, kidney stone rates vary between 4%-9%, and for women, kidney stone rates range between 2%-4%.

Previous studies dealt with the connection between sialolithiasis and nephrolithiasis were inconclusive. To the authors' best knowledge no studies were done to examine the associations between nephrolithiasis and dental calculus. Thus, the aim of this study is to compare the mineral composition of both dental calculus and nephrolithiasis and determine whether nephrolithiasis composition may be linked to the periodontal status.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with nephrolithiasis
* Over 18 years old

Exclusion Criteria:

* Pregnant woman, uncontrolled diabetes (HbA1c > 7.5%), patients who received periodontal treatment in the past 6 months, smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with kidney stone.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
the composition of both specimens | the analysis will take 9 months
  The X-ray diffraction of both kidney stone and dental calculus will result in the composition of the two, and comparison will be done

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No